CLINICAL TRIAL: NCT05344833
Title: Post-Autologous Transplant Maintenance With Isatuximab and Lenalidomide in Minimal Residual Disease Positive Multiple Myeloma
Acronym: HEME-18
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: University of Illinois at Chicago (Other)
Collaborators: Huntsman Cancer Institute (Other)
Responsible Party: Principal Investigator, Karen Sweiss, Principal Investigator, University of Illinois at Chicago
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2021-1101
Record Dates: First submitted 2022-04-19; First posted 2022-04-25 (Actual); Last update posted 2025-08-06 (Actual); Status verified 2025-05

CONDITIONS: Multiple Myeloma
MeSH Terms: conditions — Multiple Myeloma | interventions — isatuximab; Lenalidomide

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- Isatuximab and Lenalidomide Maintenance (Experimental): All participants will receive:
  Isatuximab 10mg/kg IV Days 1,8, 15, 22 Cycle 1 (all cycles 28 days). Isatuximab 10mg/kg Days 1, 15 Cylces 2 and 3. Isatuximab 10mg/kg Day 1, Cylces 4-39. Lenalidomide 10mg PO Days 1-21 Cylces 1-3 (all cycles 28 days) Lenalidomide 15mg PO Days 1-21 Cycle 4 and can continue until disease progression.
  Interventions: Drug: Isatuximab; Drug: Lenalidomide

INTERVENTIONS:
Drug: Isatuximab — Isatuximab 10mg/kg IV Days 1,8, 15, 22 Cycle 1 (all cycles 28 days). Isatuximab 10mg/kg Days 1, 15 Cylces 2 and 3. Isatuximab 10mg/kg Day 1, Cylces 4-39.
Drug: Lenalidomide — Lenalidomide 15mg PO Days 1-21 Cycle 4 and can continue until disease progression.

SUMMARY:
This is a phase II study where patients will undergo isatuximab and lenalidomide maintenance if they are MRD-positive after Autologous Stem Cell Transplant (ASCT)

DETAILED DESCRIPTION:
This is a phase II study where patients will undergo isatuximab and lenalidomide-based maintenance if they are MRD-positive after ASCT. Patients may have received equal to or less than 2 lines of induction therapy prior to ASCT. Patients will be enrolled at any time prior to ASCT or up to day 180 after ASCT.Patients will undergo disease reassessment per standard of care including BM examination and MRD testing by NGS at day 90 (+/- 30 days) of ASCT. All patients in MRD-negative (defined as 10-6) CR will be treated off study with lenalidomide monotherapy and all patients who are MRD-positive will begin treatment with isatuximab and lenalidomide, starting any time after MRD results are obtained (treatment must commence before day 180 of ASCT).Patients will be monitored for disease response and every 12 months for BM MRD status, for a total of 3 years, or until disease progression or unacceptable toxicity meeting criteria for protocol removal.

ELIGIBILITY:
NOTE: Females are considered of childbearing potential unless they are surgically sterile (have undergone a hysterectomy or bilateral oophorectomy) or they are naturally postmenopausal for at least 12 consecutive months.

12. Patients must be willing to take appropriate DVT prophylaxis, either aspirin, low molecular weight heparin, direct oral anticoagulants, or warfarin while receiving lenalidomide.

Inclusion Criteria:

1. Age > 18 years
2. Patients must have a confirmed diagnosis of multiple myeloma according to IMWG criteria. Patients with smoldering multiple myeloma, or plasma cell leukemia are not eligible. Patients must not have significant amyloid organ dysfunction per the study chair.
3. R-ISS stage 1, 2 or 3 at diagnosis. If stage at diagnosis is not known, patient may be enrolled if the intent is to treat with post -ASCT maintenance therapy.
4. Received up to or less than 2 lines of therapy prior to ASCT (as long as they did not meet IMWG refractory disease for CD38 monoclonal antibody or lenalidomide therapies as defined in exclusion).
5. Patients are planned to undergo ASCT with high dose melphalan, or have completed ASCT with high dose melphalan within the last 180 days and have not yet initiated post-ASCT maintenance.
6. Obtain at least partial response according to IMWG criteria prior to autologous stem cell transplant
7. ECOG performance status of 0, 1, or 2 within 30 days prior to enrollment.
8. Demonstrate adequate organ function as defined in the table below; all screening labs are to be obtained within 30 days prior enrollment.

   Hematologic White blood cell (WBC) ≥ 1500/mm3 Absolute Neutrophil Count (ANC) ≥ 1000/mm3 Platelets ≥ 50,000/mm3 Renal Calculated creatinine clearance ≥ 30 mL/min using either the Cockcroft-Gault formula or estimated GFR, and not requiring continuous or intermittent dialysis Hepatic Bilirubin ≤ 2.5 × upper limit of normal (ULN) Aspartate aminotransferase (AST) ≤ 2.5 × ULN Alanine aminotransferase (ALT) ≤ 2.5 × ULN Coagulation International Normalized Ratio (INR) or Prothrombin Time (PT) Activated Partial Thromboplastin Time (aPTT)1 ≤ 2 × ULN Note: Patients on anticoagulation are exempt from meeting this criterion
9. Standard of care lenalidomide will not be provided by the sponsor or study and therefore study subjects must have confirmed access to lenalidomide for use during the study at the time of enrollment.
10. Must be able to take and swallow oral medication (capsules) whole. Patients may not have any known impairment of gastrointestinal function or gastrointestinal disease that may significantly alter the absorption of study drug (e.g. ulcerative disease, uncontrolled nausea, vomiting, diarrhea, malabsorption syndrome, or small bowel resection).
11. Females of childbearing potential and males must be willing to abstain from heterosexual activity or to use 2 forms of effective methods of contraception from the time of informed consent until 5 months for females, and 1 month for males after treatment discontinuation. The two contraception methods can be comprised of two barrier methods, or a barrier method plus a hormonal method. Interventions such as IUD, tubal ligation, hormonal (birth control pills, injections, hormonal patches, vaginal rings, or implants), or partner's vasectomy, all count as one method. For women of childbearing potential (WOCBP), a second form must also be used. Men must agree to use a latex condom during sexual activity with a female of childbearing potential, irrespective of a prior vasectomy, during the study treatment and for 1 month after the end of treatment. Females of childbearing potential agree to not plan a pregnancy for 1 month after the last dose of study medication. Females of childbearing potential must agree to ongoing pregnancy testing during the treatment period.

    NOTE: Females are considered of childbearing potential unless they are surgically sterile (have undergone a hysterectomy or bilateral oophorectomy) or they are naturally postmenopausal for at least 12 consecutive months.
12. Patients must be willing to take appropriate DVT prophylaxis, either aspirin, low molecular weight heparin, direct oral anticoagulants, or warfarin while receiving lenalidomide.

Exclusion Criteria:

1. Refractory to anti-CD38 monoclonal antibody therapy OR lenalidomide as defined by the IMWG (defined as non-responsive or progressive disease on therapy or within 60 days of last treatment).
2. Prior intolerance to isatuximab or lenalidomide.
3. Prior allogeneic stem cell transplant.
4. Prior solid organ transplant requiring immunosuppressive therapy.
5. Known additional malignancy that is active and/or progressive requiring treatment; exceptions include adequately treated basal cell or squamous cell skin cancer, in situ cervical cancer, adequately treated Stage I or II cancer from which the patient is currently in complete remission, or any other cancer from which the patient has been disease free for three years.
6. Known CNS involvement by multiple myeloma, defined by positive CSF cytology for plasma cells, leptomeningeal involvement, or parenchymal CNS plasmacytoma at time of enrollment. Lumbar puncture is not required.
7. Treatment with any investigational drug within 30 days prior to enrollment.
8. Planned transplant is considered part of tandem autologous transplant approach for newly diagnosed MM.
9. Uncontrolled intercurrent illness including, but not limited to, ongoing or active infection, symptomatic congestive heart failure, unstable angina pectoris or coronary angioplasty, unstable cardiac arrhythmia (ongoing cardiac dysrhythmias of NCI Common Terminology Criteria for Adverse Events [CTCAE] v5.0 Grade ≥ 2), intracardiac defibrillators, known cardiac metastases, or abnormal cardiac valve morphology (≥ Grade 3), or known psychiatric illness/social situations that would limit compliance with study requirements.
10. Pregnant women are excluded from this study because lenalidomide is an agent with the potential for teratogenic or abortifacient effects. Because there is an unknown but potential risk for adverse events in nursing infants secondary to treatment of the mother with lenalidomide, breastfeeding should be discontinued if the mother is treated with lenalidomide.
11. Patients with known history of testing positive for human immunodeficiency virus (HIV) or known acquired immunodeficiency syndrome (AIDS) may be enrolled if the viral load by polymerase chain reaction (PCR) is undetectable with active treatment and absolute lymphocyte count ≥ 350/ul. Antiviral therapy for HIV should continue throughout the study.
12. Patients with a positive test for hepatitis B virus surface antigen (HBsAg) and/or HBV DNA indicating uncontrolled or active HBV infection. Patients with negative HBsAg and positive HBV viral load can be evaluated by a specialist for start of anti-viral therapy and study treatment can be proposed if HBV viral load becomes negative and other study criteria are met. Participants can be eligible if anti-HBc IgG is positive, but HBsAg and HBV viral load is negative (i.e., cleared infection).
13. Patients with known hepatitis C virus (HCV) viral load indicating acute or chronic infection might be enrolled if the viral load by PCR is undetectable with/without active treatment. If a patient was started on antiviral therapy prior to study enrollment, antiviral therapy should continue throughout the study.

NOTE: HIV, Hep B, and Hep C viral testing is not required and this criterion apply only to patients with a known history of HCV infection.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2023-01-05 (Actual); Primary Completion 2030-12 (Estimated); Study Completion 2030-12 (Estimated)

PRIMARY OUTCOMES:
Number of participants that have MRD-negative CR rate, defined as 10-6 | 1 year
  Evaluate the number of participants that have MRD-negative at 1 year that were MRD-positive multiple myeloma (MM) treated with isatuximab and lenalidomide based maintenance after ASCT

SECONDARY OUTCOMES:
Observed length of time of progressive free survival (PFS) | 3 years
  Number of days participants remain PFS
Observed length of time of overall survival (OS) | 3 years
  Number of days participants remain OS
Number of participants that achieve a deeper MRD-negative CR rate, defined as 10-6 | 1 year
  Evaluate the number of participants that achieve a deeper MRD-negative at 1 year that were MRD-positive in MM treated with isatuximab and lenalidomide based maintenance after ASCT
Number of participants that convert from MRD-positive to MRD-negative disease status in MM patients | 3 years
  Evaluate number of participants that convert from MRD-positive to MRD-negative disease status in MM patients receiving isatuximab and lenalidomide based maintenance
Number of participants that have an International Myeloma Working Group (IMWG) defined response rate of MM patients receiving isatuximab and lenalidomide based maintenance | 3 years
  Evaluate the number of participants that have an IMWG defined response rate
Number of participants that have MRD-negative CR rates of MM patients receiving isatuximab and lenalidomide based maintenance | 3 years
  Evaluate the number of participants that have MRD-negative CR rates
Number of occurrences of treatment-related adverse events (AE) in MM patients receiving isatuximab and lenalidomide based maintenance | 3 years
  Evaluate the number of occurrences of treatment-related AES
Evaluate health related quality of life in MM patients receiving isatuximab and lenalidomide based maintenance | 3 years
  Complete European Organization for Research and Treatment of Cancer Quality of Life Questionnaires-C30 questionnaire at 3 years. The higher the score the worse the subject's health is and the lower the score the better the subject's health is
Evaluate health related quality of life in MM patients receiving isatuximab and lenalidomide based maintenance | 3 years
  Complete European Organization for Research and Treatment of Cancer Quality of Life Questionnaires-Multiple Myeloma Module at 3 years. The higher the score the worse the subject's health is and the lower the score the better the subject's health is and the lower the score the better the subject's health is
Evaluate health related quality of life in MM patients receiving isatuximab and lenalidomide based maintenance | 3 years
  Complete European Quality of Life Five Dimensions Questionnaire-5-level at 3 years. The higher the score the worse the subject's health is and the lower the score the better the subject's health is

CONTACTS AND LOCATIONS:
Locations (1):
- University of Illinois at Chicago, Chicago, Illinois, United States